CLINICAL TRIAL: NCT00035217
Title: Follow-Up Study for Men Diagnoses With Prostate Cancer Through Participation in a Prostate Specific Antigen Screening Program
Brief Title: Follow-Up Study for Men Diagnosed With Prostate Cancer Through Participation in a Prostate Specific Antigen Screening Program
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Urological Research Foundation (Other)
Other Study IDs: NCRR-M01RR00036-0838
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
There is controversy concerning the preferred treatment for men with localized prostate cancer with regard to the relative effectiveness of different treatments in controlling the cancer and how different treatments affect the patient's quality of life. The purpose of this research is to describe the disease course of prostate cancer and to determine the effectiveness, potential complications, and quality of life after different treatments in men with prostate cancer detected via screening with prostate-specific antigen (PSA) and/or digital rectal examination

ELIGIBILITY:
Men with prostate cancer diagnosed through the PSA screening study

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States